CLINICAL TRIAL: NCT06790563
Title: Neuromodulation of the Dorsal Genital Nerve in Persistent Genital Arousal Disorder
Acronym: NemoPGAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-16221
Record Dates: First submitted 2025-01-10; First posted 2025-01-24 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2024-12

CONDITIONS: Arousal Disorders, Sexual
Keywords: Neuromodulation; Neurostimulation; Persistent Genital Arousal Disorder
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neuromodulation (Experimental): Neuromodulation every day, for 3 weeks
  Interventions: Device: Neuromodulation

INTERVENTIONS:
Device: Neuromodulation — Neuromodulation by UCon

SUMMARY:
The goal of this clinical trial is to learn if neuromodulation of the dorsal genital nerve works to treat symptoms related to Persistent Genital Arousal Disorder in women. The main questions it aims to answer are:

What is the effect of neuromodulation on PGAD symptoms in women?

Participants will:

Use a neurosimulator every day for 3 weeks. Keep a diary of their symptoms and the number of times they used the neurostimulator Fill in questionaires

ELIGIBILITY:
Inclusion Criteria:

* Women with PGAD

Exclusion Criteria:

* Women < 18 years
* Women not able to handle the neuromodulator
* Women in whom the anatomy of the genitals precludes proper electrode placement

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Symptom severity | 8 weeks
  Symptom severity on a 5-point Likert scale, filled in daily. 1 indicates no symptoms at all, 5 indicates very severe symptoms.
Neuromodulation effect | 3 weeks
  The neuromodulation effect will be assessed using a self-reported diary, where participants are prompted daily to rate their experience of symptoms in response to the question: "How do you experience your symptoms today?" Responses are recorded on a 5-point Likert scale with the following options: "No problem," "Mild," "Moderate," "Severe," or "Very severe." This dairy is quaried during the three weeks intervention period, in which the participants use the neuromodulator device daily.
Satisfaction device | At the end of the treatment, at week 8
  The consideration of using the neuromodulator device as part of their treatment, which was asked at the end of the treatment with the question "Would you like to continue using the device as part of your treatment". Following with a 'Yes' or 'No' answer.

SECONDARY OUTCOMES:
HADS | At baseline, at the end of the intervention (week 3) and at the end of post-intervention (week 8)
  Hospital Anxiety and Depression Scale, measuring the level of anxiety and depression, both scores ranging from 0 to 21:
  0-7 : no anxiety disorder or depression 8-10 : possible anxiety disorder or depression 11-21: suspected anxiety disorder or depression
PCS | At baseline, at the end of the intervention (week 3) and at the end of post-intervention (week 8)
  Pain Catestrophizing Scale. Score ranging from 0 to 52, in which a higher score indicates a higher level of pain catestrophizing.
QoL | At baseline, at the end of the intervention (week 3) and at the end of post-intervention (week 8)
  Quality of Life measured with the EQ-5D-3L (EuroQol-5 Dimensions-3 Levels). The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. Higher EQ VAS score indicated higher self-related health.
Patient Global Impression of Improvement | During follow-up (after week 8)
  Patient Global Impression of Improvement (PGI-I) is a scale to rate the patients condition now, as compared with how it was prior to before beginning treatment on a scale from 1. Very much better to 7. Very much worse.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud Unversity Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No